CLINICAL TRIAL: NCT06773767
Title: A Randomized, Two-way, Crossover, Two Parallel Groups Study to Compare the Bioavailability of 150 mg and 300 mg Trazodone Hydrochloride Tables (New Polymer) vs. 150 mg and 300 mg Trazodone Hydrochloride Contramid® Tables at Steady-state.
Brief Title: Bioavailability of Trazodone Hydrochloride (New Polymer) vs. Trazodone Hydrochloride Contramid® at Steady-state.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: SocraTec R&D GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 039(Ca)MD23341; 2024-511612-24-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-20; First posted 2025-01-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-10

CONDITIONS: Bioavailability Heathy Volunteers; Bioavailability Study; Bioequivalance
Keywords: Bioavailability; Oral multiple dose; Bioequivalence
MeSH Terms: interventions — Trazodone

STUDY DESIGN:
Intervention Model Description: To compare the bioavailability of 150 mg and 300 mg trazodone hydrochloride tablets (new polymer) vs. 150 mg and 300 mg trazodone hydrochloride Contramid® tablets at steady-state.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: 150 mg (Experimental): Treatment with two differet formulations of 150 mg trazodone hydrochloride during treatment period
  Interventions: Drug: 150 mg trazodone hydrochloride
- Group 2: 300 mg (Experimental): Treatment with two different formulations of 300 mg trazodone hydrochloride during treatment period
  Interventions: Drug: 300 mg trazodone hydrochloride

INTERVENTIONS:
Drug: 150 mg trazodone hydrochloride — To compare the bioavailability of 150 mg trazodone hydrochloride tablets (new polymer) vs. 150 mg trazodone hydrochloride Contramid® tablets at steady-state.
  Arms: Group 1: 150 mg
Drug: 300 mg trazodone hydrochloride — To compare the bioavailability of 300 mg trazodone hydrochloride tablets (new polymer) vs. 300 mg trazodone hydrochloride Contramid® tablets at steady-state
  Arms: Group 2: 300 mg

SUMMARY:
Two way, two parallel groups, crossover study to compare the bioavailability of 150 mg and 300 mg trazodone hydrochloride (new polymer) (Angelini Pharma S.p.A.) vs. 150 mg and 300 mg trazodone hydrochloride Contramid® (Angelini Pharma S.p.A.) at steady-state in 64 Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male/female
* Age: 18 to 65 years inclusive
* Body-mass index (BMI): ≥ 18.5 kg/m² and ≤ 30.0 kg/m²
* Good state of health
* Non-smoker or ex-smoker for at least 3 months
* Written informed consent (including consent on personal data processing), after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

* Existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient.
* Existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient.
* Existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient.
* Presence or history of relevant and currently treated CNS and/or psychiatric disorders.
* History of suicidal behaviour, suicidal intentions and/or suicidality among family members.
* Nurses Global Assessment of Suicide Risk (NGASR)-scale showing a high or very high risk.
* Known allergic reactions or hypersensitivity to the active ingredient used or to constituents of the pharmaceutical preparations
* History of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the Investigator
* History of alcohol intoxication
* History or known hyperthyroidism regardless of adequate treatment
* History of or known micturition disorders
* History of or known current increased intraocular pressure
* Known hypotension, orthostatic syndrome or repeated occurrence of syncope
* History of or current priapism
* History of intoxication with drugs that attenuate the CNS or antihypertensives
* Current treatment with opioids or serotonergic agents.
* Systolic blood pressure < 90 or > 139 mmHg and diastolic blood pressure < 60 or > 89 mmHg Heart rate < 50 bpm or > 90 bpm
* QTc interval > 450 ms for men and > 470 ms for women
* Laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the Investigator.
* ASAT > 20 % ULN, ALAT > 10 % ULN, bilirubin > 20% ULN and creatinine > 0.1 mg/dL ULN.
* Positive anti-HIV-test, HBs-antigen-test, or anti-HCV-test
* Vaccination against COVID-19 within the last 4 weeks prior to individual intended IMP administration
* Acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
* History of or current drug or alcohol dependence
* Positive alcohol or drug test at screening examination
* Regular intake of alcoholic food or beverages of ≥ 24 g pure ethanol for male or ≥ 12 g pure ethanol for female per day
* Subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
* Regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
* Blood donation or other blood loss of more than 400 ml within the last 6 months prior to individual enrolment of the subject
* Participation in a clinical trial with administration of any investigational medicinal product during the last 6 months prior to individual enrolment of the subject
* Simultaneous participation in another clinical trial with active ingredients
* Regular treatment with any systemically available medication
* Subjects, who report a frequent occurrence of migraine attacks
* Positive pregnancy test at screening examination
* Pregnant or lactating women
* Female subjects who do not agree to apply highly effective contraceptive methods
* Subject is vulnerable such as detained or committed to an institution by a court of law or by legal authorities or has a close affiliation with the Sponsor or the investigational site; e.g., a close relative of the investigator, dependent person, employee of the Sponsor or affiliates
* Subjects suspected or known not to follow instructions
* Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Assessment of bioequivalence of two different formulations of trazodone hydrochloride tablets 150 mg | 5 days
  Assessment of bioequivalence of Test 1 in comparison to Reference 1 after multiple dose administration under fasting conditions determined by means of the AUC(0-Tau),ss, of trazodone.
Assessment of bioequivalence of two different formulations of trazodone hydrochloride tablets 150 mg | 5 days
  Assessment of bioequivalence of Test 1 in comparison to Reference 1 after multiple dose administration under fasting conditions determined by means of the CTau, ss of trazodone.
Assessment of bioequivalence of two different formulations of trazodone hydrochloride tablets 150 mg | 5 days
  Assessment of bioequivalence of Test 1 in comparison to Reference 1 after multiple dose administration under fasting conditions determined by means of the Cmax,ss of trazodone.
Assessment of bioequivalence of two different formulations of trazodone hydrochloride tablets 300 mg | 5 days
  Assessment of bioequivalence of Test 2 in comparison to Reference 2 after multiple dose administration under fasting conditions determined by means of the AUC(0-Tau),ss of trazodone
Assessment of bioequivalence of two different formulations of trazodone hydrochloride tablets 300 mg | 5 days
  Assessment of bioequivalence of Test 2 in comparison to Reference 2 after multiple dose administration under fasting conditions determined by means of the CTau,ss of trazodone
Assessment of bioequivalence of two different formulations of trazodone hydrochloride tablets 300 mg | 5 days
  Assessment of bioequivalence of Test 2 in comparison to Reference 2 after multiple dose administration under fasting conditions determined by means of the Cmax,ss of trazodone

SECONDARY OUTCOMES:
Comparison of pharmacokinetic profiles (Concentration) of Test and Reference products | 5 days
  Concentration at the end of the dosing interval after the 1st, 2nd, 3rd and 4th IMP administration during treatment phase, considering scheduled times
Comparison of pharmacokinetic profiles (Cmin, ss) of Test and Reference products | 5 days
  Observed (absolute) minimum concentrations within the dosing interval Tau (profile day), considering scheduled times
Comparison of pharmacokinetic profiles (Fluctuation%) of Test and Reference products | 5 days
  Fluctuation as peak trough fluctuation, fluctuation% = {[Cmax,ss - Cmin,ss]/Cav} •100%
Comparison of pharmacokinetic profiles (Cav)of Test and Reference products | 5 days
  Average concentration at steady-state, Cav = AUC(0-Tau),ss/Tau
Comparison of pharmacokinetic profiles (Tmax, ss))of Test and Reference products | 5 days
  Time to reach the maximum concentration within each dosing interval (profile day), obtained directly from the data
Descriptive characterisation of safety of Test and Reference products | 8 days
  Descriptive characterisation of safety of Test and Reference products considering adverse events observed during the trial
Descriptive characterisation of tolerability of Test and Reference products | 8 days
  Descriptive characterisation of tolerability of Test and Reference products considering adverse events observed during the trial

CONTACTS AND LOCATIONS:
Locations (1):
- SocraTec R&D GmbH Clinical Pharmacology, Erfurt, Germany, Germany